CLINICAL TRIAL: NCT03419442
Title: A Retrospective, Longitudinal Multi-Center Study of Radium-223 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Multi-academic Center Study of Xofigo Patients
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19863
Record Dates: First submitted 2018-01-04; First posted 2018-02-05 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer, Castration Resistant
Keywords: Prostate cancer; Bone metastases; Xofigo
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; Docetaxel; cabazitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ra-223 therapy before chemotherapy: Treatment sequence 1 will include all mCRPC patients who received Ra-223 alone or in combination with abiraterone or enzalutamide and subsequently received chemotherapy
  Interventions: Drug: Xofigo; Drug: Taxotere; Drug: Jevtana
- Ra-223 after chemotherapy: Treatment sequence 2 includes all mCRPC patients who received chemotherapy before Radium 223 therapy
  Interventions: Drug: Xofigo; Drug: Taxotere; Drug: Jevtana

INTERVENTIONS:
Drug: Xofigo — Radium-223, 55kBq (1.49 microcurie) per kg body weight given at 4 week intervals for 6 injection
Drug: Taxotere — Docetaxel injection 75mg/m2 every 3 weeks
Drug: Jevtana — Cabazitaxel injection 25mg/m2 intravenously once every 3 weeks

SUMMARY:
The study will be conducted from a real-world perspective to describe treatment sequences involving radium-223 and chemotherapy in patients with metastatic castrate resistant prostate cancer (mCRPC) and assess overall survival (OS) associated with treatment sequences involving radium-223 and chemotherapy. While clinical trials of radium-223 has demonstrated a survival benefit in the treatment of mCRPC, both pre and post- docetaxel, study lacked exposure to second generation androgens and hence could not assess outcomes pre or post abiraterone or enzalutamide.

The specific objective of this study is to describe and compare the clinical outcomes between treatment sequences for patients with mCRPC where 1) radium-223 is used (alone or in combination with abiraterone or enzalutamide) prior to chemotherapy versus 2) radium-223 used after chemotherapy in the treatment of mCRPC. The secondary objectives are to describe the safety patterns of docetaxel use among mCRPC patients who received chemotherapy post radium-223.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one dose of radium-223 after mCRPC diagnosis
* Received at least one prescription or dose of chemotherapy for treatment of mCRPC

Exclusion Criteria:

- No documented visceral metastasis at initiation of radium-223

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of patients with CRPC and bone metastasis who have received at least one dose of radium-223 at one of the participating cancer centers. The participating centers are 4 tertiary care cancer centers (Dana Farber Cancer Institute, Tulane Cancer Center, Memorial Sloan Kettering Cancer Center and Beth Israel Deaconess Medical Center)
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 30 months
  Survival will be measured from initiation of first line therapy after mCRPC diagnosis until the date of death (from any cause).
Time to symtomatic skeletal event(SSE) | Up to 30 months
  Measured as the time from initiation of first-line therapy after mCRPC diagnosis until first SSE; for the exploratory analysis, measured as the time from initiation of radium-223 until first SSE. SSE will be identified based on the ALSYMPCA trial definition: first use of external-beam radiation therapy (EBRT) to relieve skeletal symptoms, new symptomatic pathologic vertebral or non-vertebral bone fractures, spinal cord compression, or tumor-related orthopedic surgical intervention
Reasons for treatment discontinuation | Up to 30 months
  data for treatment discontinuation for each mCRPC therapy will be collected

SECONDARY OUTCOMES:
Laboratory-based outcomes collected by questionnaire | Up to 30 months
  Data will be collected as available from initiation of docetaxel until 3 months following last dose of docetaxel
Treatments received | Up to 30 months
  measured as Yes/No
Number of hospitalizations | Up to 30 months
  along with the discharge diagnosis, as recorded in medical charts or discharge summaries
PSA PFS | Up to 30 months
  defined as death or an increase above PSA nadir by ≥25% and ≥2 ng/mL (PCWG 2008 definition for Prostate specific antigen(PSA) Progression-free survival(PFS))
Non-laboratory based clinically relevant safety outcomes | Up to 30 months
  documented in medical records
hospital length of stay | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer US, Whippany, New Jersey, United States

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/